CLINICAL TRIAL: NCT01666873
Title: Correlation Between Alignment of Lower Limb and Clinical Outcome After Total Knee Prosthesis.
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/526
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2014-12

CONDITIONS: Osteoarthritis of the Knee Joint
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- total knee prosthesis: Patients that undergo a total knee prosthesis.
  Interventions: Procedure: patients that undergo a total knee prosthesis

INTERVENTIONS:
Procedure: patients that undergo a total knee prosthesis

SUMMARY:
Evaluation of the clinical results after total knee prosthesis, and correlation with the alignment of the lower limb.

Radiological measurements by means of 3D technology will be performed. The clinical result will be stipulated by means of standardized questionnaires (KOOS, KSS and Oxford knee score-questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Patient with osteoarthritis of the knee joint, without severe bone deformation

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who have osteoarthritis of the knee joint and receive a total knee prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Clinical results after total knee prosthesis with standardized questionnaires after 6 months | 6 months after total knee prosthesis
  Standardized questionnaires (KOOS KSS en Oxford knee score-questionnaire).
Clinical results after total knee prosthesis with standardized questionnaires after 12 months. | 12 months after total knee prosthesis
  Standardized questionnaires (KOOS KSS en Oxford knee score-questionnaire).
Clinical results after total knee prosthesis with standardized questionnaires after 24 months. | 24 months after total knee prosthesis
  Standardized questionnaires (KOOS KSS en Oxford knee score-questionnaire).

SECONDARY OUTCOMES:
Alignment of lower limb, slope of lateral and medial tibial plateau, femoral slope. | 6 months after total knee prosthesis
  imaging with 3D software (MIMICS)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Victor, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be